CLINICAL TRIAL: NCT01655667
Title: Improving Diagnosis of COPD Through Characterisation of Comorbidities Present at, and Healthcare Utilisation Prior to, Diagnosis of COPD in UK. A Retrospective Primary Care Database.
Brief Title: Comorbidities and Healthcare Utilisation: Indicators for Improving COPD Diagnosis
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Department of Health, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Shuna Gould, Professor David Price, Research in Real-Life Ltd
Other Study IDs: 015/11
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Diagnosis; Primary Care; Comorbidities; Healthcare utilisation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: All patients with a coded diagnosis of COPD entered into their electronic clinical record between 1990 and 2009.

SUMMARY:
To characterise and understand the current UK COPD population including demographics, active comorbidities and missed opportunities for COPD diagnosis in the years previous to diagnosis

DETAILED DESCRIPTION:
Using real-world primary care clinical databases, ascertain whether 1) trends in respiratory resource utilisation prior to COPD diagnosis (including lower respiratory tract infections [LRTIs], consultations and hospitalisations) could be used as 'flags' to aid earlier diagnosis, and 2) characterize comorbid conditions present at the time of COPD diagnosis, and evaluate the relationship to COPD disease severity and age at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older
* Electronically coded diagnosis of COPD made between 1990 and 2009
* A minimum of three years continuous practice data including two years prior to and one year post diagnosis to ensure patients recieved COPD therapy post diagnosis
* Recieved two or more prescriptions for COPD therapies in the 12 months post diagnosis year 1.

Exclusion Criteria:

* Aged less than 40 years
* No diagnosis of COPD between 1990 and 2009
* Less than three years continuous practice data including two years prior to and one year post diagnosis
* Less than two prescriptions for COPD therapies in the 12 months post diagnosis year 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 40 years or older, with an electronically coded diagnosis of COPD made between 1990 and 2009, a minimum of three years continuous practice data including two years prior to and one year post diagnosis to ensure patients recieved COPD therapy post diagnosis (defined as two or more prescriptions for COPD therapies in the 12 months post diagnosis year 1). COPD therapies included short- and long-acting bronchodilators, inhaled corticosteroids, theophylline and leukotriene receptor antagonists.
Sampling Method: Non-Probability Sample
Enrollment: 38859 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Price, MD, Principal Investigator — Research in Real-Life Ltd; Dermot Ryan, MBBS, Study Director — University of Edinburgh; Rupert Jones, MBBS, Study Director — Peninsula College of Medinicne and Dentistry; Eric Bateman, MD, Study Director — University of Cape Town; Matt Kearney, MPH, Study Director — Department of Health, United Kingdom
Locations (1):
- Research in Real Life Ltd, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Jones RC, Price D, Ryan D, Sims EJ, von Ziegenweidt J, Mascarenhas L, Burden A, Halpin DM, Winter R, Hill S, Kearney M, Holton K, Moger A, Freeman D, Chisholm A, Bateman ED; Respiratory Effectiveness Group. Opportunities to diagnose chronic obstructive pulmonary disease in routine care in the UK: a retrospective study of a clinical cohort. Lancet Respir Med. 2014 Apr;2(4):267-76. doi: 10.1016/S2213-2600(14)70008-6. Epub 2014 Feb 13. PMID 24717623